CLINICAL TRIAL: NCT06545422
Title: Effect of St. John's Wort Oil on Skin Moisture in Intensive Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Ayşenur ÖZENÇ KOLUTEK, Nurse, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EskisehirOU-SBF-AOK-01
Record Dates: First submitted 2024-08-03; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Skin Moisture
Keywords: skin moisture; pressure ulcer; nursing; St. John's wort oil
MeSH Terms: conditions — Pressure Ulcer | interventions — Hypericum extract LI 160

STUDY DESIGN:
Intervention Model Description: Prospective pretest-posttest controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 70 experimental group patients participated in the study; St. John's wort oil was applied to the coccyx area(width 10cm, length 10cm) of the patient included in the study at the same times every day for 21 days, starting from Day 0.
  The first day of hospitalization is considered day 0 and skin moisture is measured. The skin is cleaned and dried. 4 or 5 drops of St. John's wort oil were dropped onto the area and applied with a cotton pad.The next day, skin moisture is measured then the skin is cleaned and dried and St. John's wort oil is applied again. This Process continues for 21 days and is recorded.
  Interventions: Other: St. John's wort oil
- Control Group (Other): 70 control group patients participated in the study; The skin protective barrier cream used in routine care of the coccyx region (width 10 cm, length 10 cm) of the patient included in the study was applied at the same hours every day for 21 days, starting from day 0.
  The first day of hospitalization is considered day 0 and skin moisture is measured. The skin is cleaned and dried.Barrier cream is applied to the patient's coccyx area.The next day, at the same time, skin moisture is measured, then the skin is cleaned and dried, and barrier cream is applied again.Transactions are made and recorded every day for 21 days.
  Interventions: Other: Barrier Cream

INTERVENTIONS:
Other: St. John's wort oil — To examine the effect of regularly applied St. John's Wort oil on skin moisture.
  Arms: Experimental group
Other: Barrier Cream — To examine the effect of regularly applied barrier cream on skin moisture.
  Arms: Control Group

SUMMARY:
The study was conducted to evaluate the effect of St. John's wort oil application on skin moisture in intensive care patients. The study is a prospective pre-test-post-test controlled experimental research.It has been observed that St. John's wort oil has an effect on the skin moisture of intensive care patients.

DETAILED DESCRIPTION:
Effect of St. John's Wort oil on skin moisture in intensive care patients.

The study was conducted to evaluate the effect of St. John's wort oil application on skin moisture in intensive care patients. The study is a prospective pre-test-post-test controlled experimental research.

Research data was collected at Eskisehir City Hospital, between September 1, 2023 and March 1, 2024. Descriptive Characteristics Form, Braden Risk Assessment Scale, Moisture Meter Device and St. John's wort oil were used to collect data. In the sample size power analysis of the study, the total number of samples was found to be 138 with test power ( 1-β) 0.80, α(alpha)=0.05, effect level 0.10. The research was conducted on a total of 140 patients, 70 in the experimental group and 70 in the control group. St. John's wort oil was applied to the experimental group and routine nursing care was applied to the control group for 21 days. Independent Sample t test, ANOVA (Repeated Measures test), Mann- Whitney U test, Wilcoxon test and Pearson-χ 2 cross tables were used to evaluate the data.

ELIGIBILITY:
Inclusion Criteria:

* Admission to intensive care due to internal diseases diagnosis
* The patient is immobile
* The area to be applied is determined as the Coccyx and the tissue in this area must be intact.
* No allergy to St. John's Wort oil
* No circulatory disorders in the applied area

Exclusion Criteria:

* Having a complicated diagnosis such as cancer
* Having any disease that has spread to the entire skin
* Having an allergy to topical medications or plant extracts
* The patient has different variations such as surgical operation and intensive care change (post-operative follow-up patient)
* The patient has a diagnosis of a skin disease such as dermatitis
* A wound in the coccyx area

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Experimental Group Results | Measurements were made every day from day 0 to day 20. Measurements were made every day from day 0 to day 20.
  Moisture measurement of the coccyx area was performed with a skin moisture meter.
Control Group Results | Measurements were made every day from day 0 to day 20. Measurements were made every day from day 0 to day 20.
  Moisture measurement of the coccyx area was performed with a skin moisture meter.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur ÖZENÇ KOLUTEK, researcher, Principal Investigator — student of the institution
Locations (1):
- Ayşenur ÖZENÇ KOLUTEK, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No